CLINICAL TRIAL: NCT04541017
Title: A Phase 1b/2 Study of Hu5F9-G4 (Magrolimab) in Combination With Mogamulizumab in Relapsed/Refractory Treated T-Cell Lymphoma
Brief Title: Testing the Addition of an Anti-cancer Drug, Hu5F9-G4 (Magrolimab), to the Usual Chemotherapy Treatment (Mogamulizumab) in T-Cell (a Type of Immune Cell) Lymphoma That Has Returned After Treatment or Does Not Respond to Treatment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06710; NCI-2020-06710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-203; 10384 (Other: City of Hope Comprehensive Cancer Center LAO); 10384 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2020-09-05; First posted 2020-09-09 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Mycosis Fungoides; Recurrent Mycosis Fungoides; Recurrent Mycosis Fungoides and Sezary Syndrome; Recurrent Sezary Syndrome; Refractory Mycosis Fungoides; Refractory Mycosis Fungoides and Sezary Syndrome; Refractory Sezary Syndrome; Sezary Syndrome; Stage IB Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage II Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage III Mycosis Fungoides and Sezary Syndrome AJCC v8; Stage IV Mycosis Fungoides and Sezary Syndrome AJCC v8
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — Specimen Handling; magrolimab; mogamulizumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (magrolimab, mogamulizumab), Phase Ib and Phase II (Experimental): Patients receive magrolimab IV over 2-3 hours weekly during cycles 1-2, then Q2W during cycles 3-12. Patients also receive mogamulizumab IV over at least 60 minutes weekly during cycle 1, then Q2W during cycles 2-12. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET/CT or diagnostic CT, blood sample collection, and may undergo a skin punch biopsy during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Magrolimab; Biological: Mogamulizumab; Procedure: Positron Emission Tomography; Procedure: Punch Biopsy
- Arm II (mogamulizumab), Phase II (Active Comparator): Patients receive mogamulizumab IV over at least 60 minutes weekly during cycle 1, then Q2W during cycles 2-12. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients who have received at least 2 full treatment cycles and have PD or have received at least 6 full treatment cycles and have SD may crossover to Arm I. Patients undergo PET/CT or diagnostic CT, blood sample collection, and may undergo a skin punch biopsy during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Mogamulizumab; Procedure: Positron Emission Tomography; Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT or diagnostic CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Magrolimab — Given IV
  Other Names: Hu5F9-G4; ONO 7913; ONO-7913; ONO7913
  Arms: Arm I (magrolimab, mogamulizumab), Phase Ib and Phase II
Biological: Mogamulizumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(CC Chemokine Receptor CCR4) (Human-Mouse Monoclonal KW-0761 Heavy Chain), Disulfide With Human-Mouse Monoclonal KW-0761 Kappa-Chain, Dimer; KM8761; KW 0761; KW-0761; KW0761; Mogamulizumab-kpkc; Poteligeo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Punch Biopsy — Undergo skin punch biopsy
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin

SUMMARY:
This phase Ib/II trial identifies the best dose and possible benefits and/or side effects of magrolimab when given in combination with mogamulizumab in treating patients with stage IB-IV mycosis fungoides or Sezary syndrome types of T-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Magrolimab and mogamulizumab are monoclonal antibodies that may interfere with the ability of cancer cells to grow and spread. Treatment with magrolimab in combination with mogamulizumab may stabilize cancer for longer period than the usual treatment in patients with relapsed/refractory T-cell lymphoma who have been previously treated.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and toxicity profile and to determine a safe recommended phase 2 dose (RP2D) of Hu5F9-G4 (magrolimab) when given in combination with mogamulizumab. (Phase I) II. To compare the proportion of patients who achieve a partial or complete response lasting at least 6 months (ORR6) of the combination of Hu5F9-G4 (magrolimab) and mogamulizumab versus mogamulizumab alone. (Phase II)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase I)

II. To compare the efficacy of the combination of Hu5F9-G4 (magrolimab) and mogamulizumab versus mogamulizumab alone with respect to the following endpoints (Phase II):

IIa. Overall response rate (ORR); overall response rate lasting at least 4 months (ORR4); overall response rate lasting at least 12 months (ORR12).

IIb. Duration of response (DOR). IIc. Progression-free survival (PFS). IId. Time to next treatment (TTNT).

EXPLORATORY OBJECTIVES:

I. To identify potential biomarkers that correlate with response to mogamulizumab and Hu5F9-G4 (magrolimab) including (Phase I and II):

Ia. Expression of CCR4. Ib. Somatic mutations and germline polymorphisms. Ic. Phenotyping of lymphoma and immune microenvironment. Id. Functional assay of phagocytosis.

OUTLINE: This is a phase Ib, dose de-escalation study of magrolimab followed by a phase II study. Patients in the phase Ib study receive treatment as in Arm I. Patients in the phase II study are randomized to Arm I or Arm II.

ARM I: Patients receive magrolimab intravenously (IV) over 2-3 hours weekly during cycles 1-2, then every 2 weeks (Q2W) during cycles 3-12. Patients also receive mogamulizumab IV over at least 60 minutes weekly during cycle 1, then Q2W during cycles 2-12. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET)/computed tomography (CT) or diagnostic CT, blood sample collection, and may undergo a skin punch biopsy during screening and on study.

ARM II: Patients receive mogamulizumab IV over at least 60 minutes weekly during cycle 1, then Q2W during cycles 2-12. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients who have received at least 2 full treatment cycles and have progressive disease (PD) or have received at least 6 full treatment cycles and have stable disease (SD) may crossover to Arm I. Patients undergo PET/CT or diagnostic CT, blood sample collection, and may undergo a skin punch biopsy during screening and on study.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either mycosis fungoides (MF) or Sezary syndrome (SS) by the World Health Organization (WHO) 2016 classification (Swerdlow et al., 2017), stage IB-IV by modified International Society for Cutaneous Lymphomas (ISCL)/ European Organization of Research and Treatment of Cancer (EORTC) classification (Olsen et al., 2011), without large cell transformation (LCT) at the time of screening. Patients with a history of prior LCT are permitted
* Patients must have had at least one prior course of systemic therapy
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of Hu5F9-G4 (magrolimab) in combination with mogamulizumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9.5 g/dL and transfusion independence (defined as not requiring more than 2 units of red blood cell [RBC] transfusions during the 4-week period prior to screening)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) except for subjects with Gilbert's syndrome or genetic equivalent
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 by the Cockcroft-Gault formula
* Patients must meet the following minimum wash-out window from previous treatments to the first treatment

  * >= 3 weeks for systemic anti-cancer therapies
  * >= 2 weeks for phototherapy, local radiation therapy, topical high potency corticosteroid, topical retinoid, topical nitrogen mustard, or topical toll-like receptor (TLR)-agonist
  * >= 12 weeks for total skin electron beam therapy Participants with rapidly progressive malignant disease may be enrolled prior to completion of the above periods with approval of the protocol director
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for a minimum of 3 months
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of Hu5F9-G4 (magrolimab) on the developing human fetus are unknown. For this reason and because monoclonal antibody agents as well as other therapeutic agents used in this trial (mogamulizumab) are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and continue for 4 months after the last dose of both Hu5F9-G4 (magrolimab) and mogamulizumab. Effective contraception is defined as oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide) or practice true abstinence from heterosexual intercourse. Women of childbearing potential includes any female who has experienced menarche and has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea >= 12 consecutive months). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol who are sexually active with women of childbearing potential and who have not had vasectomies must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Hu5F9-G4 (magrolimab) administration
* Female patients of childbearing potential must not be nursing or planning to be pregnant and must have a negative urine or serum pregnancy test within 30 days before randomization and within 72 hours before the first administration of study treatment

  * Female patients of childbearing potential must be willing to use one highly effective method of contraception during the study and continue for 4 months after the last dose of study treatment
  * Male patients who are sexually active with a woman of childbearing potential (WOCBP) and who have not had vasectomies must be willing to use a barrier method of contraception (condom plus spermicidal gel) and refrain from sperm donation during the study and for 4 months after the last dose of study treatment. If the partner is pregnant, male patients must use barrier method contraception (condom) during the study and for 4 months after the last dose of study treatment to prevent fetal exposure to study treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Willing to comply with clinic visit schedule and procedures including mandatory biopsies

Exclusion Criteria:

* Prior treatment with Hu5F9-G4 (magrolimab) or any agent targeting CD47-SIRPalpha
* Prior progression of disease with mogamulizumab
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and lymphopenia (any grade permitted). Residual peripheral neuropathy must have improved to grade 2 or better
* Patients who are receiving any other investigational agents
* Allogeneic hematopoietic stem cell transplant recipients with any graft-versus-host disease within the previous 3 months or requiring immunosuppression
* Active autoimmune disease that has required systemic immunosuppressive medication within the previous 3 months
* Active herpes simplex or herpes zoster. Subjects on prophylaxis for herpes who have no active signs of active infection, and whose last active infection was more than 6 months ago, may enter the study, and should continue to take the prescribed medication for the duration of the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Hu5F9-G4 (magrolimab), other monoclonal antibodies, or other agents (mogamulizumab) used in study
* Significant cardiopulmonary disease defined as

  * Acute myocardial infarction within the last 6 months
  * Unstable angina
  * Congestive heart failure New York Heart Association (NYHA) class III-IV
* Patients with uncontrolled intercurrent illness requiring antibiotics. Patients on prophylactic antibiotics for non-complicated staphylococcus colonization/infection are eligible
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are excluded
* Patients with psychiatric illness/social situations or substance abuse that would limit compliance with study requirements
* Pregnant women are excluded from this study because Hu5F9-G4 (magrolimab) is monoclonal antibody agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Hu5F9-G4 (magrolimab), breastfeeding should be discontinued if the mother is treated with Hu5F9-G4 (magrolimab). These potential risks may also apply to other agents used in this study (mogamulizumab)
* Patients with RBC transfusion dependence, defined as requiring more than 2 units of RBCs transfused during the 4-week period prior to screening. RBC transfusions are permitted during the screening period and prior to enrollment
* Patients with prior autoimmune thrombocytopenia, hemolytic anemia or Evans syndrome requiring treatment in the last 12 months
* Patients on the following medications at the time of enrollment:

  * Immunotherapy or immunosuppressive drugs (e.g. chemotherapy or systemic corticosteroids) EXCEPT for the following:

    * Intranasal, inhaled, or local steroid injection (e.g. intra-articular injection)
    * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent, if patient has been on a stable dose for at least 2 weeks prior to the first treatment
    * Low and medium potency topical corticosteroids are permitted if patient has been on a stable dose for at least 2 weeks prior to the first treatment
    * Steroids as premedication for hypersensitivity reactions (e.g. computed tomography [CT] scan premedication)
  * Growth factors (granulocyte colony stimulating factor or granulocyte macrophage colony stimulating factor) EXCEPT for erythropoietin and darbepoetin alpha
  * Herbal remedies with immunostimulating properties (e.g., mistletoe extract) or known to potentially interfere with major organ function (e.g. hypericin)
* Live vaccines are not allowed while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), typhoid (oral) vaccine, and intranasal influenza vaccines (e.g., Flu-Mist). However, seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Khodadoust, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (18):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eight patients were enrolled in the Phase Ib portion of the study. However, due to early study termination, two patients did not initiate treatment. As a result, six patients were included in the final analysis.
Period: Overall Study
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was closed following a full clinical hold issued by the FDA for magrolimab, as well as the sponsor's decision to discontinue further development of the drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [28 to 68] |  | 50 [28 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Magrolimab When Given in Combination With Mogamulizumab (Phase Ib)
Description: The phase 1b portion of the trial was designed to determine a RP2D of Hu5F9-G4 (magrolimab) and was planned to enroll 6-18 patients.
Time Frame: Up to 4 weeks from the first infusion of magrolimab (priming infusion)
Population: as for baseline characteristics
Measure: Number; unit: mg/kg
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 6 | 0
mg/kg | 30 |

2. Primary Outcome: Overall Response Rate at 6 Months (ORR6) (Phase II)
Description: Will be defined as the proportion of patients who have a partial or complete response to therapy AND a duration of response >= 6 months. Will use a stratified Cochran-Mantel-Haenszel chi-squared test to compare between-group differences in ORR6 proportion. Will also conduct a secondary analysis on the intent-to-treat population (all patients randomized to a therapy and assigned a study number) and an efficacy evaluable set (all patients who received the first 12 weeks of treatment and completed the week 12 response assessment).
Time Frame: At 6 months
Population: The Phase II portion of the study was never opened. The study was closed following a full clinical hold issued by the FDA for magrolimab, as well as the sponsor's decision to discontinue further development of the drug.
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Response Rate (ORR) (Phase Ib)
Description: Defined as the proportion of patients who have a partial or complete response to therapy as defined by the global response score.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 6 | 0
Participants | 2 |

4. Secondary Outcome: Overall Response Rate at 4 Months (ORR4) (Phase II)
Description: Will be defined as the proportion of patients who have a partial or complete response to therapy AND a duration of response >= 4 months. Will be assessed by the chi-squared method.
Time Frame: At 4 months
Population: as for outcome 2
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Response Rate at 12 Months (ORR12) (Phase II)
Description: Will be defined as the proportion of patients who have a partial or complete response to therapy AND a duration of response >= 12 months. Will be assessed by the chi-squared method.
Time Frame: At 12 months
Population: as for outcome 2
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Will be assessed by the Kaplan-Meier method and the log-rank test.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
Population: as for outcome 2
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Response (DOR) (Phase II)
Description: Will be assessed by the Kaplan-Meier method and the log-rank test.
Time Frame: From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrence or progressive disease is objectively documented, assessed up to 2 years
Population: as for outcome 2
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Next Treatment (TTNT) (Phase II)
Description: Will be assessed by the Kaplan-Meier method and the log-rank test.
Time Frame: From the start of treatment on this protocol to time of the next anti-neoplastic therapy, assessed up to 2 years
Population: as for outcome 2
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post-discontinuation of treatment, up to two years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II | Arm II (Mogamulizumab), Phase II
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II (N=6) | Arm II (Mogamulizumab), Phase II (N=0)
Fever (General disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Magrolimab, Mogamulizumab), Phase Ib and Phase II (N=6) | Arm II (Mogamulizumab), Phase II (N=0)
Anemia (Blood and lymphatic system disorders) | 2 (15) | 0 (0)
Other: Hemagglutination (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ST changes on EKG (Cardiac disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (6) | 0 (0)
Other: Muscle spasm (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (12) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (12) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (left leg swelling) (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (10) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0)
fractured tooth (General disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (8) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (28) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (9) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
RT wrist tendon repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
moderately dysplastic melanocytic nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (26) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (13) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (30) | 0 (0)
Rosacea to both cheeks (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Squamous Cell Carcinoma of RT Upper Arm (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04541017/Prot_SAP_000.pdf
  • Informed Consent Form: P10384_A07Consent(Untracked).pdf (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04541017/ICF_001.pdf
  • Informed Consent Form: P10384_A07Consent2(Untracked).pdf (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04541017/ICF_002.pdf